CLINICAL TRIAL: NCT05944848
Title: A Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of CL-197 Capsules Administered in Single Dose in Healthy Participants
Brief Title: A Study of CL-197 Capsules in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR-CL-197-101
Record Dates: First submitted 2023-07-03; First posted 2023-07-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: HIV-1
Keywords: HIV-1; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1mg group (Experimental): Single oral dose of 1 mg CL-197 capsules or CL-197 placebo
  Interventions: Drug: 1 mg CL-197 capsules
- 10mg group (Experimental): Single oral dose of 10 mg CL-197 capsules or CL-197 placebo
  Interventions: Drug: 10 mg CL-197 capsules or CL-197 placebo
- 30mg group (Experimental): Single oral dose of 30 mg CL-197 capsules or CL-197 placebo
  Interventions: Drug: 30 mg CL-197 capsules or CL-197 placebo
- 60mg group (Experimental): Single oral dose of 60 mg CL-197 capsules or CL-197 placebo
  Interventions: Drug: 60 mg CL-197 capsules or CL-197 placebo
- 100mg group (Experimental): Single oral dose of 100 mg CL-197 capsules or CL-197 placebo
  Interventions: Drug: 100 mg CL-197 capsules or CL-197 placebo

INTERVENTIONS:
Drug: 1 mg CL-197 capsules — Single oral dose of 1 mg CL-197 capsules or CL-197 placebo administered following ≥10 hour fast
  Arms: 1mg group
Drug: 10 mg CL-197 capsules or CL-197 placebo — Single oral dose of 10 mg CL-197 capsules or CL-197 placebo administered following ≥10 hour fast
  Arms: 10mg group
Drug: 30 mg CL-197 capsules or CL-197 placebo — Single oral dose of 30 mg CL-197 capsules or CL-197 placebo administered following ≥10 hour fast
  Arms: 30mg group
Drug: 60 mg CL-197 capsules or CL-197 placebo — Single oral dose of 60 mg CL-197 capsules or CL-197 placebo administered following ≥10 hour fast
  Arms: 60mg group
Drug: 100 mg CL-197 capsules or CL-197 placebo — Single oral dose of 100 mg CL-197 capsules or CL-197 placebo administered following ≥10 hour fast
  Arms: 100mg group

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetic characteristics of CL-197 capsules in health conditions.

DETAILED DESCRIPTION:
In this trial, 46 healthy participants will be enrolled, 6 healthy participants in 1mg group, 40 healthy participants distributed equally in other four groups: 10mg group, 30mg group, 60mg group and 100mg group, including thier respective placebo control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects, aged 18~45 (including boundary values), both male and female;
2. Body mass index (BMI) should be in the range of 19.0-26.0 (including the boundary value) (BMI = weight (kg) / height 2 (m2)), the body weight of male subjects should be ≥ 50.0kg, and the body weight of female subjects should be ≥ 45.0kg;
3. Those who have no family plan within 2 weeks before screening and within 3 months after the end of the trial and agree to use effective non-pharmacological contraception during the trial;
4. Understand and sign the informed consent form voluntarily.

Exclusion Criteria:

1. Allergic constitution, with a history of drug or food allergies, especially allergic to any ingredient in this product and excipients;
2. Those with a history of hypoglycemia in the past;
3. Pre-test medical history, physical examination, laboratory items and test-related examinations and abnormal tests have clinical significance, and the clinical research doctor judges to be unqualified;
4. Those with a history of smoking in the 12 months before screening (the number of cigarettes per day≥ 5);
5. Those who have a history of alcoholism in the 12 months before screening (drink ≥ 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 150mL of wine) or positive alcohol breath test (test value>0mg/100mL) before enrollment;
6. Those who have a history of drug abuse within 12 months before screening or who have tested positive for addictive substances before enrollment;
7. Those who have undergone surgery within 3 months before screening, especially those who have undergone surgery that will affect drug absorption, distribution, metabolism, and excretion, or those who plan to undergo surgery during the study;
8. Any drugs that interact with investigational drugs, such as potent CYP3A inhibitors (such as clarithromycin, indinavir, itraconazole, etc.), have been used within 30 days before screening;
9. Have a previous history of cardiovascular, hepatic, renal, lung, digestive tract, nerve and other diseases, especially any surgical condition or condition that may affect the absorption, distribution, metabolism and excretion of drugs, or any surgical condition or condition that may pose a hazard to the subjects participating in the trial;
10. Those who have a febrile illness within 3 days before screening;
11. Those who have participated in other clinical trials within 3 months before screening;
12. Those who have a history of taking any prescription drugs, over-the-counter drugs, Chinese herbal medicines, and health products within 14 days before screening;
13. Those who consumed excessive tea, coffee and/or beverages rich in caffeine, xanthine and alcohol (more than 8 cups, 1 cup = 250mL) every day within 3 months before screening;
14. Those who have lost blood or donated blood ≥ 200mL within 8 weeks before screening;
15. Pregnant and lactating women;
16. Those who cannot tolerate venipuncture blood collection and/or have a history of blood sickness and needle sickness;
17. Those who have been vaccinated against the new coronavirus within 1 week before screening, or those who have received other vaccines within 3 months before screening;
18. Those who are not considered suitable to enter this test by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
The Safety and Tolerability of CL-197 Capsules ：Incidence of Treatment-Emergent Adverse Events as Assessed by The NCI CTCAE V5.0 Grading Criteria | Up to 29 days post-dose
  The degree of adverse events observed in the trial would be determined by the NCI CTCAE v5.0 grading criteria, and the adverse events related to the test drug (definitely related, likely to be related, and possibly related) would be terminated in the following cases, and the previous dose would be used as the MTD of the single-dose tolerance test.

SECONDARY OUTCOMES:
The Peak Plasma Concentration (Cmax) of CL-197 Capsules | Up to 672 hours post-dose in 30mg group and 60 mg group; Up to 162 hours post-dose in other groups
  The index components in human blood samples would be measured by LC-MS/MS, and the peak plasma concentration (Cmax) would be calculated.
The Area Under the Plasma Concentration Versus Time Curve (AUC) of CL-197 Capsules | Up to 672 hours post-dose in 30mg group and 60 mg group; Up to 162 hours post-dose in other groups
  The index components in human blood samples would be measured by LC-MS/MS, and the area under the plasma concentration versus time curve (AUC) would be calculated.
The Elimination Half-Life (t1/2) of CL-197 Capsules | Up to 672 hours post-dose in 30mg group and 60 mg group; Up to 162 hours post-dose in other groups
  The index components in human blood samples would be measured by LC-MS/MS, and the elimination half-life (t1/2) would be calculated.
The Accumulate Urinary Drug Excretion (Ae) of CL-197 Capsules | Up to 672 hours post-dose in 30mg group and 60 mg group; Up to 162 hours post-dose in other groups
  The index components in human urine samples would be measured by LC-MS/MS, and the accumulate urinary drug excretion (Ae) would be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Fusheng, Principal Investigator — Medical Director
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China